CLINICAL TRIAL: NCT00112996
Title: Prevention of Cisplatin- or Oxaliplatin-Induced Peripheral Neuropathy With Alpha-Lipoic Acid: A Placebo-Controlled Phase III Trial
Brief Title: Alpha-Lipoic Acid in Preventing Peripheral Neuropathy in Patients Receiving Chemotherapy for Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CDR0000403155; MDA-CCC-0327; MDA-2004-0728; 2004-0728 (Other: UT MD Anderson Cancer Center); NCI-2009-00636 (Registry Identifier: NCI CTRP); 3U10CA045809-15S1 (NIH); NCT00705029 (obsolete NCT alias)
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Neurotoxicity; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: neurotoxicity; unspecified adult solid tumor, protocol specific; unspecified childhood solid tumor, protocol specific
MeSH Terms: conditions — Neurotoxicity Syndromes | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I: Alpha-Lipoic Acid (Experimental): Oral alpha-lipoic acid three times daily for at least 24 weeks in the absence of unacceptable toxicity.
  Interventions: Drug: alpha-lipoic acid
- Arm II: Placebo (Placebo Comparator): Oral placebo three times daily for at least 24 weeks in the absence of unacceptable toxicity.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: alpha-lipoic acid — Oral two 300 mg ALA sustained release tablets initiated 4 days after last dose of platinum and discontinued 2 days before next scheduled platinum dose, continued for 24 weeks.
  Arms: Arm I: Alpha-Lipoic Acid
Other: placebo — Given orally two similar color and sized placebo control tablets three times a day continued for 24 weeks.
  Arms: Arm II: Placebo

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Chemoprotective drugs, such as alpha-lipoic acid, may protect normal cells from the side effects of chemotherapy. Alpha-lipoic acid may also prevent damage to nerves that carry information to and from the brain and spinal cord to the rest of the body. It is not known whether alpha-lipoic acid is more effective than placebo in preventing peripheral neuropathy.

PURPOSE: This randomized phase III trial is studying alpha-lipoic acid to see how well it works compared to placebo in preventing peripheral neuropathy in patients receiving chemotherapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare whether treatment with alpha-lipoic acid vs placebo decreases the severity and frequency of peripheral neuropathy in cancer patients receiving a cisplatin- or oxaliplatin-containing chemotherapy regimen.
* Compare the protective effect duration of these drugs in these patients.

Secondary

* Determine large sensory fiber integrity associated with platinum-induced peripheral neuropathy, as measured by three timed functional tests comprising fastening 6-buttons, walking 50 feet, and placing coins in a cup, in patients treated with these drugs.
* Compare the number of chemotherapy courses and doses received by patients treated with these drugs.

Tertiary

* Compare the optimal tumor response (disease progression, stable disease, partial response, or complete response) to chemotherapy in patients treated with these drugs.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to prior platinum-containing treatment (yes vs no). Patients who received prior treatment are further stratified according to prior cumulative platinum exposure (cisplatin < 200 mg/m^2 or oxaliplatin < 750 mg/m^2 vs cisplatin 200-399 mg/m^2 or oxaliplatin 750-999 mg/m^2 vs cisplatin >400 mg/m^2 or oxaliplatin > 1,000 mg/m^2). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral alpha-lipoic acid* three times daily for at least 24 weeks in the absence of unacceptable toxicity.
* Arm II: Patients receive oral placebo* three times daily for at least 24 weeks in the absence of unacceptable toxicity.

NOTE: *In both arms, patients begin taking study drug 4 days after completion of each chemotherapy treatment and continue taking study drug until 2 days before their next scheduled chemotherapy treatment.

Patients' symptoms of peripheral neuropathy, pain, and functional tests are assessed at baseline and then at weeks 6-8, 12, 24, 36, and 48.

PROJECTED ACCRUAL: A total of 244 patients (122 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Scheduled to receive a cisplatin- or oxaliplatin-containing chemotherapy regimen for cancer
* No established clinical neuropathy
* No clinically evident CNS metastases, including leptomeningeal metastases

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin < 2 mg/dL

Renal

* Creatinine < 2 mg/dL OR
* Creatinine clearance > 45 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must have a normal state of arousal
* No confusion or memory or concentration deficit
* No history of diabetes mellitus requiring oral medication or insulin treatment
* No chronic alcoholism
* No other active central nervous system (CNS) disease (e.g., dementia or encephalopathy)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No carboplatin, vincristine, vinblastine, paclitaxel, or docetaxel for 6 months prior, during, and 6 months after study treatment

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Concurrent medications that can modify peripheral neuropathy (e.g., gabapentin, lamotrigine, carbamazepine, phenytoin, or tricyclic antidepressants) are allowed provided there is no dose adjustment within 2 weeks before study entry and during study participation
* No concurrent vitamin E (including multivitamins that contain vitamin E) ≥ 100 IU per day
* No concurrent physical modality (e.g., anodyne [monochromatic near-infrared photoenergy, 890 nm], microcurrent, or transcutaneous electrical neural stimulation) for peripheral neuropathy related symptoms unless physical or occupational therapy for functional training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2007-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Severity of neuropathy | Up to 48 weeks
  Severity of neuropathy as measured by the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity Questionnaire total score at baseline and at 6-8, 12, 24, 36, and 48 weeks

SECONDARY OUTCOMES:
Group Differences in Change scores | Up to 48 weeks
  Group differences in change scores from baseline at 6-8, 12, 24, 36, and 48 weeks
Number of courses received | Up 48 weeks
Optimal tumor response | Up to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ying Guo, MD, MS, Principal Investigator — M.D. Anderson Cancer Center
Locations (13):
- United States (13):
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Horizon Oncology Center, Lafayette, Indiana
  - CCOP - Wichita, Wichita, Kansas
  - Cabrini Center for Cancer Care at Christus St. Frances Cabrini Hospital, Alexandria, Louisiana
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - CCOP - Greenville, Greenville, South Carolina
  - University of Texas M.D. Anderson CCOP Research Base, Houston, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org